CLINICAL TRIAL: NCT05912036
Title: The CORTEX Project: a Pre-post Randomized Controlled Feasibility Trial Evaluating the Efficacy of a Computerized COgnitive Remediation ThErapy Progeam for Adult Inpatients With anoreXia Nervosa
Brief Title: The CORTEX Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03C214
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Cognitive remediation therapy; Randomized controlled trial; Cognitive flexibility; Motivation to change; Quality of life
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: CRT involves the completion by patients of a series of tasks on a computer while a trained facilitator engages them in a discussion about the tasks. Patients are encouraged to verbalize their process and to do self-check-ins to gauge their performance
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CA-CRT (Experimental): Computer-Assisted Cognitive Remediation Therapy
  Interventions: Behavioral: CRT
- TAU (No Intervention): Treatment as Usual

INTERVENTIONS:
Behavioral: CRT — CA-CRT treatment will entail exercises aimed to improve cognitive strategies, encourage subjects' reflection on their way of thinking, and explore the possibility of implementing new schemas in everyday life. The CA-CRT program will employ a range of cognitive exercises and tasks to address cognitive inflexibility and weak central coherence. The treatment will consist of 10 individual CA-CRT sessions, 2 times per week for 5 weeks, for a duration of 40 minutes per session with 15 individual CA-CRT sessions, 3 times a week for 5 weeks, with a duration of 30 minutes per session
  Arms: CA-CRT

SUMMARY:
Background: This study aims to evaluate the feasibility and efficacy of a novel Computer-Assisted Cognitive Remediation Therapy (CA-CRT) program as adjunctive treatment to standard care (TAU) in improving cognitive skills in adult inpatients with anorexia nervosa (AN) Methods: A multicenter randomized controlled trial (RCT) will be conducted to compare the experimental condition with controls receiving TAU only. A minimum sample of 54 subjects with a diagnosis of AN will be recruited in each site. After the initial screening, participants will be randomized to either the experimental group or the control condition. The treatment will last 5 weeks and consists of 10 individual CRT sessions with 15 individual CA-CRT sessions. The impact of the intervention on selected primary and secondary outcomes will be tested at the end of the intervention.

Expected results: We expect subjects assigned to the CA-CRT group to develop more flexible and holistic thinking styles, and achieving increased clinical outcomes.

DETAILED DESCRIPTION:
For this reason, the present multicenter Randomized Control Trial (RCT) aims to implement a new CA-CRT for AN (CA-CRT-AN) and to test its feasibility and efficacy as an adjunctive intervention on selected neuropsychological (cognitive flexibility, verbal fluency, visuospatial processing, and attention) and psychological measures (eating disorders, health-related quality of life - HRQoL, and motivation to change) in populations of inpatients with AN following a nutritional rehabilitation program compared to controls following the treatment already used in the clinics (TAU).

Patients with AN will be invited to take part in the study at admission to each rehabilitation center according to the above-mentioned inclusion/exclusion criteria, and those eligible will be randomly assigned to either the experimental (CA-CRT) or control group (TAU).

Before the randomization, they will be asked to sign the informed consent to participate in the research and complete the psychodiagnostic (BAI, BDI II, OCI-R) and psychological (EDE-Q, WHOQOL-BREF, URICA) measures under the supervision of a clinical psychologist independent of the study. The selected neuropsychological measures will be also administered at baseline Randomization will be stratified by center and performed using permuted block technique within each site by a researcher independent of the study. Subjects will be assigned to one of two conditions: both groups received usual hospital care, and the experimental group, in addition, will receive the CA-CRT treatment.

At the end of the treatment (after 5 weeks), subjects in both conditions will be re-administered with neuropsychological tests and psychological measures The total duration of the research will be 6 months, considering a discontinuous enrollment related to the admission to the clinics

ELIGIBILITY:
Inclusion criteria for the participants in the study will be: (1) receiving a diagnosis of AN according to DSM 5 criteria (American Psychiatric Association, 2013) following psychiatric evaluation; (2) being over 18 years; (3) having Italian citizenship; (4) signing the informed consent to participate in the study.

Participants will be excluded from the study if: (1) having specific learning disabilities (SLDs), (2) having intellectual disability, psychosis, previous head injury, history of psychotropic substance use, or other clinical conditions (e.g., visual impairment, hearing impairment; etc.) that would prevent them from following the intervention Subjects will not be excluded if already receiving psychopharmacological therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
mental flexibility (ability to change rule sets), and problem-solving skills | pre-pos intervention (5 weeks)
  Wisconsin Card Sorting Test

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Castelnuovo, Principal Investigator — IRCCS Istituto Auxologico

IPD SHARING:
Plan to Share IPD: Undecided
Under request